CLINICAL TRIAL: NCT00832598
Title: 18F] FACBC and [18F] FLT PET Imaging in Central Nervous System Tumors
Brief Title: [18F] FACBC and [18F] FLT PET Imaging in Central Nervous System Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-142
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-02

CONDITIONS: Brain Cancer; Gliomas
Keywords: 18F-FACBC; PET scan imaging; 08-142
MeSH Terms: conditions — Brain Neoplasms; Glioma

ARMS (1):
- PET imaging (Experimental): We will perform [18F]FACBC PET and [18F]FLT PET imaging on 30 patients with gliomas scheduled for treatment with pathway inhibitor agents such as receptor tyrosine kinase inhibitors, antibodies (e.g., bevacizumab), VEGF-Trap, etc.
  Interventions: Radiation: [18F]FACBC PET and [18F]FLT PET imaging

INTERVENTIONS:
Radiation: [18F]FACBC PET and [18F]FLT PET imaging — [18F]FACBC PET and [18F]FLT PET imaging on 30 patients with gliomas scheduled for treatment with pathway inhibitor agents such as receptor tyrosine kinase inhibitors, antibodies (e.g., bevacizumab), VEGF-Trap, etc. Patients with measurable disease on MRI will undergo PET imaging at baseline (prior-to) and after approximately 1 month of treatment.

SUMMARY:
The purpose of this study is to help us understand gliomas, one type of brain tumor. This research protocol makes pictures of gliomas. We will take pictures of the glioma before and after treatment. The pictures are made with a positron emission tomography (PET) scanner. PET scans use radioactive markers to "see" cancer cells. We plan to use two different radioactive markers, [18F]FACBC and [18F]FLT, to "see" if the glioma responds to the treatment being recommended by the doctor. We are investigating whether one or both of these types of PET scans can help us to better understand gliomas and their response to treatment.

We expect these pictures will give us information the your tumor and may help us to understand why the treatment that the patient is receiving is affecting the tumor the way that it is. We also hope to collect information about the amount of radioactivity exposure. We will measure radioactivity exposure to the tumor, brain and other organs.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC.
* Child-bearing age females must be non-pregnant,(documented by a negative pregnancy test within the last 2 weeks), non-lactating, and must be using adequate contraception or be surgically sterile.
* Patients with gliomas
* Patients planning to start anti-AKT and/or anti-VEGF directed therapies .
* Patients with measurable disease on MRI or CT neuroimaging.

Exclusion Criteria:

* Patient is incontinent of urine or stool (which would make them unable to tolerate lying still for 60 minutes).
* Patient cannot tolerate lying still for a 60 minute session in the PET tomograph.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Blasberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- PET Imaging: We will perform [18F]FACBC PET and [18F]FLT PET imaging on participants with gliomas scheduled for treatment with pathway inhibitor agents such as receptor tyrosine kinase inhibitors, antibodies (e.g., bevacizumab), VEGF-Trap, etc.
Period: Overall Study
Arm/Group | PET Imaging
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PET Imaging
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 46 [34 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Determine & Comp Biodistribution, Clearance, & Dosimetry of [18F]FACBC & [18F]FLT Tissue/Organs w/i the Field of View of the Dynamic PET Imag Studies prior-to & During Anti-AKT &/or Anti-VEGF Directed Therapies Alone or in Combin With Radia for Glioma.
Time Frame: 2 years
Population: Data was not collected
Arm/Group | PET Imaging
Number analyzed (Participants) | 0

2. Secondary Outcome: Compare [18F]FACBC PET & [18F]FLT PET Results With MRI Imaging in Patients With Recurrent Gliomas (n=30).
Time Frame: 2 years
Population: Data was not collected
Arm/Group | PET Imaging
Number analyzed (Participants) | 0

3. Secondary Outcome: Explore if [18F]FACBC PET and [18F]FLT PET Imaging Can be Related to Molecular Markers (AKT, VEGFR, and Related Signaling/Biologic Changes by Immunohistochemistry and/or Analysis of Flash Frozen Tissue)
Time Frame: 2 years
Population: Data was not collected
Arm/Group | PET Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | PET Imaging
All-Cause Mortality (participants affected / at risk) | 12/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET Imaging (N=13)
Confusion (Psychiatric disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Memory-impairment (Nervous system disorders) | 1
Pain - headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT00832598/Prot_SAP_000.pdf